CLINICAL TRIAL: NCT06083727
Title: Primary Cesarean Section in Primigravida and Muligravida in Sohag and Al Balyana Cities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sahar Nasser Fathy, resident at obstetric and gynacology department at sohag university hospial, Sohag University
Other Study IDs: Soh-Med-23-09-03MS
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Primary Cesarean Section

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- primigravida
  Interventions: Other: rate of cesarean section
- multigravida
  Interventions: Other: rate of cesarean section

INTERVENTIONS:
Other: rate of cesarean section — rate of primary cesarean section in primigravida and multigravida

SUMMARY:
cesarean section and vaginal delivery are two methods of delivery, cesarean section somtimes indicated for obstetrical reason but primary cesarean section especially in primigravida might have a preference of the mode of delivery

ELIGIBILITY:
Inclusion Criteria:

* all primigravida with gestational age more than 28 weeks and above who have come for delivery
* multigravida upto gravida 4 with gestational age more than 28 weeks and above who has had one previous viable vaginal delivery
* women between 18 and 45 years

Exclusion Criteria:

* primigravida women <28 weeks
* multigravida <28 weeks
* patient having previous history of myomectomy or hystrotomy
* gravida 5 and more

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: all primigravida with gestational age more than 28 weeks and above who have come for delivery
  * multigravida upto gravida 4 with gestational age more than 28 weeks and above who has had one previous viable vaginal delivery
  * women between 18 and 45 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2024-03-24 (Estimated); Study Completion 2024-03-24 (Estimated)

PRIMARY OUTCOMES:
rate | 6 months
  rate of primary cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided